CLINICAL TRIAL: NCT06928155
Title: Feasibility and Usability of Immersive Virtual Reality for People With Dependency
Brief Title: Inclusive Rehabilitation: Virtual Reality as a Tool to Improve the Quality of Life of Dependent Persons
Acronym: REVIVIR
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad de Almeria (Other)
Responsible Party: Principal Investigator, Raul Romero-del Rey, Ph.D., Universidad de Almeria
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: TRFE-SI-2024/005
Record Dates: First submitted 2025-04-07; First posted 2025-04-15 (Actual); Last update posted 2025-07-29 (Actual); Status verified 2025-07

CONDITIONS: People With Dependency
Keywords: quality of life, dependency, virtual reality, rehabilitation
MeSH Terms: interventions — Smart Glasses; Exercise; Resistance Training

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): The intervention group will receive immersive virtual reality sessions twice a week, for a total of 6 weeks, with sessions lasting no more than 30 minutes.
  Interventions: Device: Immersive Virtual Reality with Head Mounted Display
- Control group (Active Comparator): The control group will continue with their usual physiotherapy treatment, which includes aerobic exercises and strength training.
  Interventions: Other: Aerobic exercise and strength training

INTERVENTIONS:
Device: Immersive Virtual Reality with Head Mounted Display — The intervention will be carried out with an immersive virtual reality device, specifically, with a head mounted display. Specifically, it is the "MetaQuest 3" model.
  Arms: Intervention group
Other: Aerobic exercise and strength training — The combination of aerobic and strength training is part of the conventional physiotherapy treatment carried out at the center.
  Arms: Control group

SUMMARY:
The project explores the use of virtual reality (VR) as a tool to improve the quality of life of people with dependence, providing immersive and personalized environments that support physical, neurological and psychological rehabilitation. VR makes it possible to practice complex movements, improve strength and coordination, reduce stress and anxiety, and enhance brain plasticity through adapted simulations that are also motivating and safe for users. This approach facilitates more effective rehabilitation than traditional therapies by allowing repetition and visualization of movements that are difficult to perform in real life. The El Saliente Association, in collaboration with the University of Almeria, leads this initiative that seeks to promote the autonomy, inclusion and emotional well-being of people with dependence. With specific objectives such as improving motor function, stimulating neuroplasticity, reducing pain through immersive distraction and enhancing independence, the project uses VR sessions in controlled environments. In addition, activities that simulate everyday situations will be designed to facilitate the transfer of acquired skills to the real environment. The work plan is divided into design, development, implementation and analysis phases, including participant selection, software development, pilot testing and evaluation of results. At each stage, data will be collected to measure the effectiveness of the intervention, with the ultimate goal of publishing the findings in scientific forums and replicating the experience in other contexts. Day center facilities and a residential complex will provide the necessary spaces and materials to carry out the interventions. Expected outcomes include increased motivation and adherence to therapy, faster functional recovery and an overall improvement in quality of life, including increased self-esteem and reduced anxiety. This project promises a significant advance in the use of technology for inclusive rehabilitation, with benefits not only for patients but also for the advancement of innovative therapeutic solutions in the field of dependency.

DETAILED DESCRIPTION:
The world's population is aging rapidly. Globally, the number of people aged 80 years and older is projected to more than triple between 2017 and 2050, from 137 million to 425 million (1). Various studies have shown that the four most common health conditions in older adults are decreased motor skills, increased obesity, cognitive impairment, and psychological disorders, leading to lower quality of life (2, 3).

To combat this challenge, several emerging assistive technologies that improve quality of life in older populations have been explored, including Internet-based physical activity programs, gamification to improve physical activity [4], etc. Virtual reality (VR) is also an emerging technology with the potential to improve well-being and quality of life [5], muscle activity and balance, and physical activity [6], with evidence of beneficial effects on social, emotional states, and cognition [7].

VR offers a highly personalized virtual environment that allows exercises to be tailored to the specific needs of each patient. Users can practice movements in realistic and motivating scenarios, which increases their engagement and motivation during rehabilitation sessions. By allowing complex, customized movements to be simulated, VR facilitates the visualization and repeated practice of actions that, in the physical world, would be difficult or impossible to execute. This constant repetition stimulates the neural pathways associated with movements, promoting neuroplasticity and improving coordination and muscle strength.

Therefore, the purpose of this study is to describe the impact of the application of Immersive Virtual Reality on the mobility and anxiety levels of the participants, as well as to explain adherence, the presence of adverse effects and the usability of this tool.

ELIGIBILITY:
Inclusion Criteria:

* Over 18 years of age
* Patients who agree to participate in the study and sign the informed consent form.

Exclusion Criteria:

* Those with severe visual impairment, vertigo, epilepsy or psychosis, and who may interfere with the normal performance of interactive voice response (IVR) tasks, will be excluded as a precaution.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 172 (Estimated)
Dates: Start 2025-06-01 (Actual); Primary Completion 2025-10-28 (Estimated); Study Completion 2025-12-28 (Estimated)

PRIMARY OUTCOMES:
Anxiety levels | At baseline, at 6 weeks and at 2 months.
  Anxiety levels will be measured using the Generalized Anxiety Disorder (GAD-7).

SECONDARY OUTCOMES:
Adherence levels | At baseline, at 6 weeks and at 2 months
  The level of adherence to the intervention will be measured by keeping a record of users who do or do not complete the sessions, in order to establish the dropout rate.
Functional mobility | At baseline, at 6 weeks and at 2 months
  Functional mobility will include the evaluation of gait and balance using the Tinetti scale (0-28 points).
Ability to perform activities of daily living | At baseline, at 6 weeks and at 2 months
  The ability to perform activities of daily living will be measured using the Barthel Index (0-100 points).
Cognitive impairment | At baseline, at 6 weeks and at 2 months
  Cognitive impairment will be measured using the Lobo Mini Cognitive Test.
Usability/Acceptability | At 6 weeks and at 2 months
  The usability or acceptability of the intervention will be measured with the Usability Scales System (SUS).
Feasibility/cybersickness | At 6 weeks and at 2 months.
  The feasibility of the intervention will be measured according to the occurrence of adverse symptomatology associated with the use of virtual reality. For this purpose, the "Simulator Sickness Questionnaire" (SSQ) will be used.

CONTACTS AND LOCATIONS:
Locations (1):
- Asociación "El Saliente", Almería, Andalusia, Spain

IPD SHARING:
Plan to Share IPD: No